CLINICAL TRIAL: NCT04095494
Title: Study Of the Nitrous Oxide Perception in Health Students
Acronym: SONOPS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UK
Record Dates: First submitted 2019-08-30; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-08

CONDITIONS: Nitrous Oxide Abuse
Keywords: EMONO; Health students

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Nitrous oxide use — In order to evaluate the perception of the Nantes health students we wish to place an anonymous survey concerning their training, their knowledge of the legislative framework governing the use of EMONO and their personal and professional experience around nitrous oxide.

SUMMARY:
In order to evaluate the perception of the Nantes health students we wish to place an anonymous survey concerning their training, their knowledge of the legislative framework governing the use of EMONO and their personal and professional experience around nitrous oxide.

DETAILED DESCRIPTION:
The use of nitrous oxide in the form of EMONO (Equimolar Mixture of Nitrous Oxide and Oxygen) is common practice in the medical field in France since obtaining the AMM in France in 2001. It is used daily in the hospital services for its analgesic and anxiolytic properties in order to obtain a conscious sedation of the patient during the realization of painful care. Its use in liberal practice has been authorized since 2009 in France following the confirmation of its security by clinical studies.

In its medical use, the use of nitrous oxide is subject to numerous regulations; EMONO's various presentations are on the I list of poisonous substances and are subject in part to the regulation of narcotics (secure storage, obligation to report flights ...) in France. The use of this substance can only be done under medical prescription, in adapted premises, by a medical or paramedical staff specifically trained, and whose knowledge will be periodically reevaluated. All conditions of use and storage of EMONO are specified in the French Code of Public Health (Article L5123-2) and, since it is authorized in a non-hospital environment, enhanced monitoring of pharmacovigilance and addictovigilance and a Risk Management Plan (RMP) has been put in place.

Paradoxically, apart from the supervised medical use, it is very simple to obtain nitrous oxide. It is found in particular in whipped cream cartridges in a pure concentration (100% N2O) over-the-counter and unregulated. In this form it is transferred into balloons by consumers in order to be inhaled. Also known as laughing gas, it is diverted from its original use for its euphoric properties and its effects (visual and sensory distortions) that last only a few minutes.

The regulations governing the use of nitrous oxide have been put in place because the toxicity of the latter is recognized in particular during chronic use. The risks associated with the acute consumption of nitrous oxide are essentially hypoxia with even cases of death recorded in the literature. Nitrous oxide consumed chronically can inactivate vitamin B12 by oxidizing its cobalt ion causing neurological pathologies (myoneuropathies).

The risks related to nitrous oxide are certainly rare but known. The fact that it can be easily obtained gives this "legal drug" a special status combining rare but existing side effects and the risk of public abuse.

The medical and paramedical professions are the more at risk populations as the use of this molecule becomes more popular. In the literature, the death cases mainly concern dentists for exemple.

The use of nitrous oxide in the form of EMONO is not necessarily part of the core curriculum of medical and paramedical education but today requires specific training. However, all health students will one day be brought to use it in the realization of painful care. It is fundamental to respect the defined framework of this drug use so as not to end up in a situation of abuse (on the part of patients as well as that of practitioners).

There is the question of student training. Is the initial medical training on nitrous oxide sufficient? Do students have a fair perception of this medicine as well as its use and misuse? In order to evaluate the perception of the students we wish to place an anonymous questionnaire concerning their training, their knowledge of the legislative framework governing the use of MEOPA and their personal and professional experience around nitrous oxide.

ELIGIBILITY:
Inclusion Criteria:

* Being an health students in Nantes University

Exclusion Criteria:

* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is that of healthy students in Nantes who are exposed to the use of EMONO and their personal and professional experience with nitrous oxide.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
nitrous oxide use in the form of EMONO | 5 minutes
  Investigate the percentage of health students who had contact with EMONO Survey on the use of EMONO among health students

CONTACTS AND LOCATIONS:
Overall Officials: Tony Prud'homme, Principal Investigator — Nantes University Hospital
Locations (1):
- Chu de Nantes, Nantes, France